CLINICAL TRIAL: NCT05928520
Title: Comparison of Analgesic Efficacy of Topical Tramadol Versus Topical Lidocaine in the Control of Post Operative Pain in Children After Tonsillectomy
Brief Title: Pain Management in Pediatric Adenotonsillectomy
Acronym: AZU
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Abdelwahab Saleh, Professor of Anesthesia, Intensive Care, and Pain Management, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Alazhar University
Record Dates: First submitted 2023-06-01; First posted 2023-07-03 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Pain Management
Keywords: Topical analgesia; Lidocaine; Tramadol; Modified Visual Analogue Scale
MeSH Terms: conditions — Agnosia | interventions — Tramadol; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tramadol group (Experimental): Swabs soaked with tramadol 5% 2 mg/kg diluted with saline 0.9%
  Interventions: Drug: Tramadol 5%; Drug: Lidocaine 2%
- Lidocaine group (Active Comparator): Swabs soaked with lidocaine 2% 2mg /kg diluted with saline 0.9%
  Interventions: Drug: Tramadol 5%; Drug: Lidocaine 2%

INTERVENTIONS:
Drug: Tramadol 5% — Topical tramadol 5%
  Other Names: Topical tramadol
Drug: Lidocaine 2% — Topical Lidocaine 2%
  Other Names: Topical Lidocaine

SUMMARY:
Tonsillectomy is considered one of the most frequent minor surgeries conducted on a day-case basis on children, and usually associated with pain and sore throat. This study aimed to include 80 children, ASA physical status I&II aged 4-15 years, and undergoing tonsillectomy. The purpose of this study is to determine the analgesic efficacy of topically applied lidocaine and tramadol in relieving post-operative pain in children following tonsillectomy.

DETAILED DESCRIPTION:
Pain and sore throat following tonsillectomy are typical. As a result, the issue of adequate post-tonsillectomy pain management remains a significant therapeutic obstacle. Several medications, including nonsteroidal anti-inflammatory drugs, corticosteroids and narcotics have been utilised to alleviate pain following tonsillectomy. Nevertheless, they have numerous undesirable negative consequences. NSAIDs may impede hemostasis and increase the propensity for bleeding. Opioid may result in respiratory depression, nausea, and vomiting. Consequently, the major purpose of this study is pain alleviation with minimal adverse effects.

This prospective, randomized, double-blind controlled clinical study will include 80 children, undergoing tonsillectomy, to receive either topical tramadol 5% or lidocaine 2%. Modified Visual Analogue Scale (m-VAS), bleeding, nausea, vomiting, sore throat, otalgia, fever, halitosis, and constipation will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent acute tonsillitis
* Chronic tonsillitis
* Tonsillar hypertrophy with or without obstructive sleep apnea

Exclusion Criteria:

* Parent refusal
* Hypersensitivity
* History of bronchial asthma
* Renal impairment
* Impaired liver function
* Bleeding disorders

Ages: 4 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
modified visual analogue pain score (m-VAS) | "day 7" after surgery
  It is 0-10 scale, color-coded (blue to red) scale. The scale also included depictions of faces, from happy to sad. Zero indicates no pain, 1-3 indicates mild pain, 4-7 indicates moderate pain, and 8-10 indicates severe agony.

SECONDARY OUTCOMES:
Post-tonsillectomy bleeding | Within 7 days after surgery
  Percentage of cases
Postoperative nausea and vomiting | Within 7 days after surgery
  Percentage of cases
Halitosis | Within 7 days after surgery
  Percentage of cases
Otalgia | Within 7 days after surgery
  Percentage of cases
Fever | Within 7 days after surgery
  Percentage of cases
Trismus | Within 7 days after surgery
  Percentage of cases
Time to first ibuprofen rescue analgesia | Within 7 days after surgery
  The time from the end of the surgical procedure to the first request of ibuprofen in minutes
Time to first oral fluid intake | Within the first day after surgery
  It is measured in hours, beginning from the end of the procedure
Time to first oral solid intake | Within the first day after surgery
  It is measured in hours, beginning from the end of the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Abdelwahab Saleh, Principal Investigator — Faculty of Medicine, AlAzhar University

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data will be available indefinitely following publication. Data related to the study protocol, informed consent, clinical study report and the statistical analysis plan will be available to anyone who wishes to access the data.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately following publication and no end date.
Access Criteria: Data will be available indefinitely following publication. Documents will be allowed for sharing through email. A third party will decide the quality and type of data requests. The criteria for reviewing requests based on the quality of the requests.

REFERENCES:
- [Background] Mitchell RB, Archer SM, Ishman SL, Rosenfeld RM, Coles S, Finestone SA, Friedman NR, Giordano T, Hildrew DM, Kim TW, Lloyd RM, Parikh SR, Shulman ST, Walner DL, Walsh SA, Nnacheta LC. Clinical Practice Guideline: Tonsillectomy in Children (Update)-Executive Summary. Otolaryngol Head Neck Surg. 2019 Feb;160(2):187-205. doi: 10.1177/0194599818807917. PMID 30921525
- [Background] Aldamluji N, Burgess A, Pogatzki-Zahn E, Raeder J, Beloeil H; PROSPECT Working Group collaborators*. PROSPECT guideline for tonsillectomy: systematic review and procedure-specific postoperative pain management recommendations. Anaesthesia. 2021 Jul;76(7):947-961. doi: 10.1111/anae.15299. Epub 2020 Nov 17. PMID 33201518